CLINICAL TRIAL: NCT02148406
Title: Programs to Support You During Chemotherapy (Pro-You): Feasibility
Brief Title: Programs to Support You During Chemotherapy (Pro-You)
Acronym: Pro-You
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stephanie Sohl, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VICC GI 1416; NCI-2014-00905 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICC GI 1416 (Other: Vanderbilt-Ingram Cancer Center); P30CA068485 (NIH)
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Depressive Symptoms; Fatigue; Psychosocial Effects of Cancer and Its Treatment; Stage IIA Colon Cancer; Stage IIA Rectal Cancer; Stage IIB Colon Cancer; Stage IIB Rectal Cancer; Stage IIC Colon Cancer; Stage IIC Rectal Cancer; Stage IIIA Colon Cancer; Stage IIIA Rectal Cancer; Stage IIIB Colon Cancer; Stage IIIB Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
Keywords: Yoga; Mind-body therapies; Fatigue; Colorectal cancer; Depressive symptoms
MeSH Terms: conditions — Depression; Fatigue; Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — Yoga; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (YST intervention) (Experimental): Patients undergo YST intervention comprising four individualized, 30 minute in-person sessions that instructs skills to enhance mindfulness and promote relaxation during outpatient chemotherapy sessions in weeks 2, 4, 6, and 8. Patients practice awareness - noticing the current state and establishing relaxed breathing for 5 minutes; movement - 7 minutes of gentle movements coordinated with the breath (such as raising and lowering the arms); breathing practice - 3 minutes of inhaling cool air as if through a straw; and meditation - 5 minutes of focus on letting go of physical and mental tension. Patients review a handout describing the YST and to encourage patients to practice daily with strategies to increase adherence to home practice. Patients also receive an audio recording of the YST and devices to play the recording and are asked to keep a home practice log.
  Interventions: Behavioral: Yoga Skills Training (YST); Other: questionnaire administration; Other: fatigue and depressive symptom assessment and management; Other: psychological stress assessment; Other: laboratory biomarker analysis
- Arm II (attention control) (Active Comparator): Patients attend four 30-minute sessions with an interventionist in weeks 2, 4, 6, and 8. During these sessions, patients are encouraged to discuss their experiences while receiving chemotherapy and do not receive instruction of movement, meditation or breathing practices. Patients will also be asked to write brief diary entries daily at home.
  Interventions: Other: questionnaire administration; Other: fatigue and depressive symptom assessment and management; Other: psychological stress assessment; Other: laboratory biomarker analysis; Other: Attention Control

INTERVENTIONS:
Behavioral: Yoga Skills Training (YST) — Undergo YST
  Other Names: yoga
  Arms: Arm I (YST intervention)
Other: questionnaire administration — Ancillary studies
Other: fatigue and depressive symptom assessment and management — Ancillary studies
  Other Names: fatigue and depressive assessment/management
Other: psychological stress assessment — Ancillary studies
Other: laboratory biomarker analysis — Correlative studies
Other: Attention Control
  Arms: Arm II (attention control)

SUMMARY:
This randomized pilot clinical trial studies Yoga Skills Training or attention control in reducing fatigue and depressive symptoms during chemotherapy in patients with stage II-IV colorectal cancer. Yoga Skills Training consists of meditation, movement and breathing practices that aim to promote mindfulness and relaxation. Attention control consists of conversations with a caring professional with a recommendation to complete daily home diaries. It is not yet known whether Yoga Skills Training is better than attention control at reducing fatigue and depressive symptoms in patients undergoing chemotherapy.The purpose of this initial feasibility study is to refine study procedures.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain preliminary data on the efficacy of the Yoga Skills Training (YST) for improving the targeted outcomes (primary: fatigue; secondary: depressive symptoms) as compared to the attention control (AC).

II. To explore potential mediators (psychological stress, circadian disruption, inflammation) and moderators (gender, dose of the YST, outcome expectancies) of the effects of the YST on targeted outcomes.

III. To qualitatively assess perceived efficacy of the interventions and acceptance of daily measurement through semi-structured interviews in a subset of participants.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (YST intervention): Patients undergo YST intervention comprising four individualized, 30 minute in-person sessions that instructs skills to enhance mindfulness and promote relaxation during outpatient chemotherapy sessions in weeks 2, 4, 6, and 8. Patients practice awareness - noticing the current state and establishing relaxed breathing for 5 minutes; movement - 7 minutes of gentle movements coordinated with the breath (such as raising and lowering the arms); breathing practice - 3 minutes of inhaling cool air as if through a straw; and meditation - 5 minutes of focus on letting go of physical and mental tension. Patients are given a handout describing the YST and audio recording with devices to play the recording to encourage patients to practice daily. Strategies to increase adherence to home practice will be implemented and patients will be asked to keep home practice logs.

ARM II (attention control): Patients attend four 30-minute in-person sessions with an interventionist in weeks 2, 4, 6, and 8. During these sessions, patients are encouraged to discuss their experiences while receiving chemotherapy and do not receive instruction of movement, meditation or breathing practices. Patients will also be asked to write brief diary entries daily at home.

After completion of study, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to receive first-line intravenous chemotherapy treatment for colorectal cancer (stages II-IV)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Ability to understand and the willingness to sign an informed consent document written in English

Exclusion Criteria:

* Regularly engaged (>= 3 days/week) in moderate physical activity of any kind (e.g., yoga) over the past 4 weeks
* Has a self-reported history of diagnosed sleep disorders (e.g., obstructive sleep apnea, insomnia), comorbidities associated with poor sleep or fatigue (e.g., chronic fatigue syndrome), or a job with night shifts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes in fatigue (recalled) | at 10 weeks
  Patient-Reported Outcomes Measurement Graphical and descriptive summaries of the patterns over time of these summary statistics for each of these groups will comprise a key initial phase of the analyses. Bootstrapping methods will be used to generate 95% confidence intervals for all sample descriptive statistics and effect estimates. Key statistical tests will involve between group differences in mean values and group differences in the patterns (i.e., slopes) of individual changes from respective baseline values. Evaluated using mixed-effects (or multilevel) generalized linear modeling procedures with robust variance estimation.

SECONDARY OUTCOMES:
Changes in depressive symptoms (recalled and daily) | Baseline up to 14 weeks
  Graphical and descriptive summaries of the patterns over time of these summary statistics for each of these groups will comprise a key initial phase of the analyses. Bootstrapping methods will be used to generate 95% confidence intervals for all sample descriptive statistics and effect estimates. Key statistical tests will involve between group differences in mean values and group differences in the patterns (i.e., slopes) of individual changes from respective baseline values. Evaluated using mixed-effects (or multilevel) generalized linear modeling procedures with robust variance estimation.
Changes in daily fatigue | Baseline up to 14 weeks
  Patient-Reported Outcomes Measurement Graphical and descriptive summaries of the patterns over time of these summary statistics for each of these groups will comprise a key initial phase of the analyses. Bootstrapping methods will be used to generate 95% confidence intervals for all sample descriptive statistics and effect estimates. Key statistical tests will involve between group differences in mean values and group differences in the patterns (i.e., slopes) of individual changes from respective baseline values. Evaluated using mixed-effects (or multilevel) generalized linear modeling procedures with robust variance estimation.
Changes in psychological stress (daily and recalled) as assessed by Perceived Stress Scale (PSS) | Baseline up to 14 weeks
  Graphical and descriptive summaries of the patterns over time of these summary statistics for each of these groups will comprise a key initial phase of the analyses. Bootstrapping methods will be used to generate 95% confidence intervals for all sample descriptive statistics and effect estimates. Key statistical tests will involve between group differences in mean values and group differences in the patterns (i.e., slopes) of individual changes from respective baseline values. Evaluated using mixed-effects (or multilevel) generalized linear modeling procedures with robust variance estimation.
Regulation of psychological stress (daily and recalled) as assessed by Positive and Negative Affect Schedule-Expanded Form and Cancer Behavior Inventory | Up to 14 weeks
  Graphical and descriptive summaries of the patterns over time of these summary statistics for each of these groups will comprise a key initial phase of the analyses. Bootstrapping methods will be used to generate 95% confidence intervals for all sample descriptive statistics and effect estimates. Key statistical tests will involve between group differences in mean values and group differences in the patterns (i.e., slopes) of individual changes from respective baseline values. Evaluated using mixed-effects (or multilevel) generalized linear modeling procedures with robust variance estimation.

OTHER OUTCOMES:
Rates of home practice as assessed by daily paper logs | Up to 10 weeks
  Mean levels of rates (%s) will be assessed
Rates of survey compliance | Up to 10 weeks
  Mean levels of rates (%s) will be assessed
Rates of efficacy expectations as assessed by adapted items the Life Orientation Test-Revised | Up to 10 weeks
  Mean levels of rates (%s) will be assessed
Rates of satisfaction | Up to 14 weeks
  Mean levels of rates (%s) will be assessed.
Reliability of the responses | Up to 14 weeks
Changes in circadian disruption (daily and recalled) as assessed by actigraphy and the Godin's Leisure Score Index | Baseline up to 14 weeks
  Graphical and descriptive summaries of the patterns over time of these summary statistics for each of these groups will comprise a key initial phase of the analyses. Bootstrapping methods will be used to generate 95% confidence intervals for all sample descriptive statistics and effect estimates. Key statistical tests will involve between group differences in mean values and group differences in the patterns (i.e., slopes) of individual changes from respective baseline values. Evaluated using mixed-effects (or multilevel) generalized linear modeling procedures with robust variance estimation

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sohl, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/